CLINICAL TRIAL: NCT04798053
Title: Impact of COVID-19 Pandemic and Social Distancing on Mental Health of Chronic Inflammatory Rheumatism Affected Patients
Acronym: EMOPTION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Societe Francaise de Rhumatologie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2020/36
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-03

CONDITIONS: Covid19; Rheumatic Fever; Mental Disorder
Keywords: Covid19; chronic inflammatory rheumatism; stress; Patient reported outcomes
MeSH Terms: conditions — COVID-19; Rheumatic Fever; Mental Disorders | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient affected by a chronic inflammatory rheumatism (Experimental): patient affected by a chronic inflammatory rheumatism (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, Systemic lupus, Still disease, scleroderma…),
  Interventions: Behavioral: Questionnaire; Biological: blood sample and salivary sample
- Controls (Active Comparator): patient affected by a non-inflammatory or degenerative musculo-skeletal disease during the containment period
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — 14-item Perceived Stress Scale (PSS-14), 9-item Patient Health Questionnaire (PHQ-9 questionnaire), State Trait Inventory Anxiety questionnaire (STAI questionnaire), Post-traumatic Stress Disorder Checklist Scale (PCL-S questionnaire)
Biological: blood sample and salivary sample — 10 ml whole blood for Peripheral blood and 2 ml saliva sample. Only for 100 cases.
  Arms: Patient affected by a chronic inflammatory rheumatism

SUMMARY:
Recent studies have highlighted the consequences of COVID-19 pandemic and social distancing on mental health of individuals. The aim of this study is to evaluate those consequences within a sample of inflammatory chronic rheumatism affected patients, taking into account the well-known key role of stress in the set-up of such diseases.

DETAILED DESCRIPTION:
The previous H1N1 and SRAS-1 pandemics, that required to containment and quarantine, have lead to the emergence of mental symptoms such as stress, anxiety, insomnia… The French COCONEL study during the COVID pandemic have shown the major psychological impact of this crisis on the population, leading to stress and fears.

Stressful life events are well-known factors of chronic inflammatory rheumatisms set-up or flare. The aim of this study is therefore to evaluate the psychological impact of COVID-19 pandemic on chronic inflammatory rheumatism (CIR) affected patients.

A case-control prospective multicentric study will be performed on 212 CIR patients versus 106 controls to compare the stress level in each group. Patient reported outcomes will be evaluated, using electronic questionnaires, as well as classical clinical informations on CIR evolution during a 6-months follow-up period. An ancillary study on 100 patients will also be realized to quantify cytokine serum levels and determinate transcriptomic profiles.

ELIGIBILITY:
For the cases:

Inclusion Criteria:

* adult patient (age over 18 years old)
* patient affected by a chronic inflammatory rheumatism (rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, Systemic lupus, Still disease, scleroderma…)
* patient without any language difficulty
* affiliated to an health insurance system
* and who agree to participate in the study

For controls :

Inclusion Criteria:

* adult patient (age over 18 years ol
* patient affected by a non-inflammatory or degenerative musculo-skeletal disease during the containment period,
* patient without any language difficulty,
* affiliated to an health insurance system,
* and who agree to participate in the study.

For cases and controls :

Exclusion Criteria:

* pregnant or lactating patient
* psychiatric patient
* patient under guardianship or other legal protection regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 259 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-12-09 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline stress level according to 10-item Perceived Stress Scale (PSS-10) at 3 months and 6 months after inclusion | At inclusion (day 0), 3 months and 6 months after inclusion
  that varies between 10 and 50 with higher values mean greater difficulties to deal with stress

SECONDARY OUTCOMES:
Proportion of patients affected by depression according to 9-item Patient Health Questionnaire (PHQ-9) | At inclusion (day 0), 3 months and 6 months after inclusion
  that varies between 0 and 27 with higher values mean greater severity of depression
Proportion of patients affected by anxiety symptoms according to State-Trait Anxiety Inventory questionnaire | At inclusion (day 0), 3 months and 6 months after inclusion
  that varies between 20 and 80 with higher values mean higher levels of anxiety
Proportion of patients affected by post-traumatic stress disorder symptoms according to Post-traumatic stress disorder Check-List Scale (PCL-S) questionnaire | At inclusion (day 0), 3 months and 6 months after inclusion
  that varies between 17 and 85 with higher values mean greater intensity of stress disorder
Evaluation of tobacco consumption evolution compared to the pre-COVID19 pandemic (less, same or more) | At inclusion (day 0), 3 months and 6 months after inclusion
Evaluation of alcohol consumption evolution compared to the pre-COVID19 pandemic (less, same or more) | At inclusion (day 0), 3 months and 6 months after inclusion
Evaluation of drugs consumption evolution compared to the pre-COVID19 pandemic (less, same or more) | At inclusion (day 0), 3 months and 6 months after inclusion
Evaluation of CIR treatments compliance continuation compared to the pre-COVID19 pandemic (without any modification, intensification, diminution, discontinuation). | At inclusion (day 0), 3 months and 6 months after inclusion
Evaluation of chronic inflammatory rheumatism activity scores using Visual Analog Scale (VAS) | At inclusion (day 0), 3 months and 6 months after inclusion
  that varies between 0 and 100mm with higher value mean higher value means higher level of disease activity.
Evaluation of the impact of COVID-19 diagnostic on the stress level according to 10-item Perceived Stress Scale (PSS-10) | At inclusion (day 0), 3 months and 6 months after inclusion
  that varies between 10 and 50 with higher values mean greater difficulties to deal with stress
Evaluation of the impact of COVID-19 diagnostic on CIR activity using Visual Analog Scale (VAS) | At inclusion (day 0), 3 months and 6 months after inclusion
  that varies between 0 and 100mm with higher value mean higher value means higher level of disease activity
Levels of pro-inflammatory cytokines in sera of CIR patients | At inclusion (day 0) and 6 months after inclusion
  TNF-alpha, IL1, IL6, IL10, IL12, IL17, TGF-beta), expressed in UI per milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: Thierry SCHAEVERBEKE, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (7):
- France (7):
  - CHU de Bordeaux - service de rhumatologie, Bordeaux
  - AP-HP - Hopital Henri Mondor - service de rhumatologie, Créteil
  - CHRU de Lille - Service de rhumatologie, Lille
  - CHU de Montpellier - service de rhumatologie, Montpellier
  - AP-HP - Hopital Cochin - service de rhumatologie, Paris
  - CHU de Saint-Etienne - service de rhumatologie, Saint-Etienne
  - CHU de Toulouse - service de rhumatologie, Toulouse